CLINICAL TRIAL: NCT04151641
Title: Evaluation of Absorption and Metabolism of Phenolic Compounds From Mangoselect®, an Extract of Mangosteen. Comparison of Two Versions During a Randomized, Double-blinded and Cross-over Trial
Brief Title: Mangoselect®: Characterization, Pharmacokinetics and Bioavailability of Xanthone Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: MNGBDP
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Dietary Supplement: MNGDPF; Dietary Supplement: MNGEF
- Sequence 2 (Experimental)
  Interventions: Dietary Supplement: MNGDPF; Dietary Supplement: MNGEF

INTERVENTIONS:
Dietary Supplement: MNGDPF — Standardized mangosteen extract in dry powder form
Dietary Supplement: MNGEF — Standardized mangosteen extract in encapsulated form

SUMMARY:
The aim of this study is to compare pharmacokinetics and bioavailability of phenolic compounds, mainly xanthones, from a mangosteen extract, either ingested in a dry powder form or in an encapsulated form. Absorption and metabolism will be determined by measuring urinary excretion of phenolic metabolites and blood metabolic profile over 72 hours by means of High Pressure Liquid Chromatography (HPLC) coupled with tandem mass spectroscopy.

The design of this study is a cross-over, double-blind and randomized trial on 10 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent study
* Stated willingness to comply with all the study procedures and availability for the duration of the study
* Male and female
* Normal BMI range (18.50-24.99)
* In good general health as evidenced by medical history
* Ability to take oral medication and be willing to adhere to lifestyle considerations

Exclusion Criteria:

* Current use of any medication or food supplement
* Pregnancy or lactation
* Known allergic reaction to mangosteen
* Metabolic disorders or any kind of disease
* Currant smoker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Difference in urinary metabolites excretion between MNGDPF (Mangoselect dry powder form) and MNGEF (Mangoselect encapsulated form) | Baseline (post-ingestion), 0-3 hours, 3-6 hours, 6-10 hours, 10-14 hours, 14-24 hours, 24-48 hours, 48-72 hours
  Urine samples will be collected in baseline and up to 72h after ingestion of the supplement according to the time frame. Urinary metabolites will be identified and quantified by High Pressure Liquid Chromatography-Mass spectrometry (HPLC-MS).

SECONDARY OUTCOMES:
Difference in plasma concentration of phenolic metabolites between MNGDPF and MNGEF | Baseline (post-ingestion), 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 19 hours, 24 hours, 48 hours
  Plasma samples will be collected in baseline and up to 48h after ingestion of the supplement according to the time frame. Plasma metabolites will be identified and quantified by HPLC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz, Principal Investigator — UCAM
Locations (1):
- UCAM, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No